CLINICAL TRIAL: NCT03843827
Title: Randomized Comparative Study Between Classic Laryngeal Mask Airway and I Gel Airway in Obese Patients Having BMI 35-40 During Elective Non Abdominal Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: N 34-2017/Ms
Record Dates: First submitted 2019-02-08; First posted 2019-02-18 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: LMA Vs I Gel
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: Investigators hypothesize that both supraglottic devices, the classic LMA and i gel are effective in ventilation of obese patient.
Who Masked: Participant, Care Provider
Masking Description: 50Patients are randomly divided by computer designed lists and then concealed in closed envelopes into 2 equal groups:
  1. Group A (n = 25), in which classic LMA is used for ventilation.
  2. Group B (n = 25), in which I gel is used for ventilation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (LMA Group) (Active Comparator): Active Comparator: Group A (LMA Group) LMA-Classic™ laryngeal mask airway (Classic™LMA) by Dr. Archie Brain into clinical practice in 1988 brought about a revolution in anesthesia. In the literature, there are over 2,500 studies supporting Classic™ LMA usage. Following the success and popularity of Classic™ LMA, many different variants of this device have been designed and marketed,trying to offer a simple and effective alternative to the endotracheal intubation.
  Interventions: Device: Laryngeal Mask Airway
- Group B (I gel Group) (Active Comparator): I gel is a new type of laryngeal mask and doesn't have an inflatable cuff. Because of its thermoplastic elastomer structure, it exactly adapts to the supraglottic tissue by binding with body temperature,thus minimising air leakage
  Interventions: Device: I gel Airway

INTERVENTIONS:
Device: Laryngeal Mask Airway — The aim of this study is to compare between cLMA and I gel regarding insertion success rate, the time of insertion, leaking pressure, assessment of position by fiber optic, hemodynamic, Spo2 for each device during insertion and maintenance of general anaesthesia and postoperative complications in obese patients
  Arms: Group A (LMA Group)
Device: I gel Airway — I gel is a new type of laryngeal mask and doesn't have an inflatable cuff. Because of its thermoplastic elastomer structure, it exactly adapts to the supraglottic tissue by binding with body temperature, thus minimising air leakage
  Arms: Group B (I gel Group)

SUMMARY:
Invistigators study both supraglottic airway devices; the classic LMA and the I GEL mask are satisfactory devices providing high airway leaking pressures. Although both devices provide high airway leaking pressures, Invistigators study revealed that the I gel mask provides a better seal with the glottic aperture and shorter time of insertion than cLMA. Both devices showed also effective ventilation, more hemodynamic stability and no episode of hypoxia with minimal post-operative complications.

DETAILED DESCRIPTION:
Because of the advantages of supraglottic devices over the conventional endotracheal intubation, they are now widely used in ventilation. The classic LMA is a first generation simple airway tube consists of two parts, the tube and the cuffed peri-laryngeal sealer mask which is designed to provide an oval seal around the laryngeal inlet. It is made of medical grade silicone; it can be autoclaved and reused many times. I gel is a new type of laryngeal mask and doesn't have an inflatable cuff. Because of its thermoplastic elastomer structure, it exactly adapts to the supraglottic tissue by binding with body temperature, thus minimising air leakage. The aim of this study is to compare between cLMA and I gel regarding insertion success rate, the time of insertion, leaking pressure, assessment of position by fiber optic, hemodynamic, Spo2 for each device during insertion and maintenance of general anaesthesia and postoperative complications in obese patients. This study was conducted in Kasr Al-Ainy Teaching Hospital, after obtaining approval from Kasr Al-Ainy hospital research ethical committee, written informed consents were taken from 50 patients, all of whom completed this study. Patients were randomly allocated into 2 equal groups, 25 each, according to the inclusion and exclusion criteria.

* GA (n=25) in which classic laryngeal mask was used for ventilation.
* GB (n=25) in which I gel was used for ventilation. In our study the median insertion time was in I gel lesser than cLMA (9 s vs 10 s) respectively that was statistically significant but clinically insignificance. Higher leaking pressure was in I gel group (25cmh2o vs 18cmh2o) than cLMA group that was statistically significant. Our main finding in the study was that both supraglottic airway devices; the classic LMA and the I GEL mask are satisfactory devices providing high airway leaking pressures. Although both devices provide high airway leaking pressures, our study revealed that the I gel mask provides a better seal with the glottic aperture and shorter time of insertion than cLMA. Both devices showed also effective ventilation, more hemodynamic stability and no episode of hypoxia with minimal postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy ASA II patients
2. both genders
3. BMI 35-40
4. aged 18 - 60 years
5. Mallampati grade I, II with airway score < 4 according to El Ganzouri score during elective non abdominal surgery ≤ 2hour e.g diagnostic arthroscopy, hysteroscopy and cataract

Exclusion Criteria:

1. ASA class III or IV
2. Age >60 years or <18 years,
3. people with hypertension, diabetes, pregnancy, gastro oesophageal reflux disease, cardiovascular ,renal disease4. difficult mask ventilation , obstructive sleep apnea ,any position rather than supine , airway score ≥ 4 according to El Ganzouri score

5. any form of sore throat ,patients allergic to any drugs used in the study 6. PCV mode if measured tidal volume was lesser than 6 ml/kg it will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Time of insertion of each device . | Half an hour
  Invistigators study Time of insertion of each device,Laryngeal Mask Airway and I gel

SECONDARY OUTCOMES:
Leaking pressure of each device. | Half an hour
  Invistigators study Leaking pressure of each device,Laryngeal Mask Airway and I gel
Confirmation of position by fiber optic | Half an hour
  Invistigators study Confirmation of position by fiber optic of each device,Laryngeal Mask Airway and I gel
Blood Pressure | 24 hours
  Investigators recorded a baseline reading of systolic blood pressure and diastolic blood pressure before insertion of both devices. A second reading was taken after insertion of both devices, just before removal. The fourth reading was recorded 1 min after removal of both devices.
Heart Rate | 24 hours
  Investigators recorded a baseline reading of heart rate, before insertion of both devices. A second reading was taken after insertion of both devices, just before removal. The fourth reading was recorded 1 min after removal of both devices.
Oxygen saturation | 24 hours
  Investigators recorded a baseline reading of Oxygen saturation before insertion of both devices. A second reading was taken after insertion of both devices, just before removal. The fourth reading was recorded 1 min after removal of both devices.
Postoperative complications | 24 hours
  With regard to postoperative complications, after removal of the device, post operative blood stain in laryngeal mask and I gel

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Not Now